CLINICAL TRIAL: NCT04328896
Title: Telemedicine Monitoring of Nocturnal Incidents of Treatment-Requiring Hypoglycemia in Older Adults With Type 1 Diabetes Miletus - A Feasibility Study
Brief Title: Telemedicine Monitoring of Nocturnal Incidents
Acronym: TELE-MONITOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Anne Peters, Professor of Clinical Medicine, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TELE-MONITOR
Record Dates: First submitted 2020-03-25; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 1; Hypoglycemia
Keywords: Remote Daily Monitoring; Continuous Glucose Monitoring; Tele-Medicine
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Intervention Model Description: This study is a 14 week, single center, pilot study of 10 subjects 65-75 yrs old with type 1 diabetes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Tele-CGM-monitoring: Subjects are remotely monitored daily through a continuous glucose monitoring (CGM) system (Dexcom G5/6) that communicates via smart phone to a Tidepool designed dashboard. Alerts set for: ≥4 hours without CGM signal, ≥2 hours 54-70 mg/dl, and 15 minutes <54 mg/dl. Tidepool dashboard automatically emails daily alerts to the Certified Diabetes Educator (CDE). If alerts occurred, the CDE performed telemedicine outreach based on type of alert.
  Interventions: Other: CGM-Tele-monitoring

INTERVENTIONS:
Other: CGM-Tele-monitoring — Baseline Visit-Visit 0
  1. Obtain informed consent
  2. Administer questionnaires
  3. Measure A1C
  4. Start study Dexcom CGM device (those already on CGM will change to the study device).
  5. The patient will be signed into Tidepool using a research code name and email.
  Visit 1-2 weeks
  1. 14 days worth of data will be downloaded from the patient's CGM device.
  2. Systems will be checked to be sure they are functioning
  3. Remote monitoring program will be activated.
  4. Telemedicine procedure will be discussed with patient; emergency contact numbers will be obtained in case patient cannot be reached
  Visit 2-14 weeks
  1. Administer questionnaires
  2. Measure A1C.
  3. Collect CGM data and compare to baseline
  Testing and Assessments:
  * Continuous glucose monitoring
  * Tidepool cloud upload
  * HbA1c
  * T1D REDEEM diabetes distress questionnaire
  * Hypoglycemia Fear Survey
  * Assessment of Severe Hypoglycemia and Diabetic Ketoacidosis

SUMMARY:
Reducing hypoglycemia is an important aspect of management of type 1 diabetes (T1D) in older adults, many of whom have hypoglycemic unawareness, cognitive impairment, or both. Continuous Glucose Monitoring (CGM) offers the opportunity to reduce hypoglycemia and its related complications such as fractures from falls and hospitalizations and improve QOL including reducing hypoglycemic fear and diabetes distress. The potential benefit of CGM in reducing hypoglycemia in the older adult population has not been well studied. Prior and on-going trials compare CGM to self-monitoring of blood glucose levels, but none look at remote daily monitoring of CGM data or provision of telemedicine based on clinic notification of hypoglycemic events. This study is a 14 week, single center, pilot study of 10 subjects 65-75 yrs old with type 1 diabetes. The primary aim is to determine the effect of continuous remote CGM reporting coupled with a telemedicine intervention (Tele-CGM program) on rates of hypoglycemia in adults with T1D >65 years old. Study staff will review Tidepool uploads and call/email to the patient if one of the following occur has occurred in the past 24 hours: ≥4 hours without CGM signal, ≥2 hours 54 - 70 mg/dl and/or 15 minutes <54 mg/dl. Tele-monitoring call will include questions to find out why the event happened and then suggestions on how to trouble shoot to avoid issues in the future. As this is a feasibility study, statistical considerations were not used.

DETAILED DESCRIPTION:
SUMMARY OF STUDY RATIONAL - Reducing hypoglycemia is an important aspect of management of T1D in older adults, many of whom have hypoglycemic unawareness, cognitive impairment, or both. CGM offers the opportunity to reduce hypoglycemia and its related complications such as fractures from falls and hospitalizations and improve QOL including reducing hypoglycemic fear and diabetes distress. Despite these potential benefits, CGM is used by only a small proportion of older adults with T1D (19% in the T1D Exchange registry). Previous studies assessing CGM efficacy have included only a small number of adults ≥ 60 years of age, excluded patients most prone to severe hypoglycemia (SH), focused on improving HbA1c rather than hypoglycemia, and used older generation CGM sensors. These studies are not generalizable to the population of older adults with T1D. The potential benefit of CGM in reducing hypoglycemia in the older adult population has not been well studied. Prior and on-going trials compare CGM to self-monitoring of blood glucose levels, but none look at remote daily monitoring of CGM data. Moreover, in none of the studies is education standardized. The follow-up of patients is done only at routine clinic visits, without any particular oversight of glucose values on an on-going basis. In some cases individual patients may share their data with a family member, but these are generally not trained medical personnel and the Dexcom provided by Medicare has the "share" feature disabled.

INTERVENTION Baseline Visit: Participants will sign informed consent, complete questionnaires, measure HbA1C, start new CGM sensor and be signed in to the Tidepool application for TeleMonitoring.

Visit 1- will occur at Week @ 2 where 14 days of CGM data will be downloaded from participants' device, systems will be checked for functioning status, remote monitoring program will be activated, telemedicine procedure will be discussed with patient; emergency contact numbers will be obtained in case patient cannot be reached.

TeleMonitoring -This will consist of an out going call/email to the patient if one of the following occur has occurred in the past 24 hours: ≥4 hours without CGM signal, ≥2 hours 54 - 70 mg/dl and/or 15 minutes <54 mg/dl. The study coordinator will be alerted each morning though the Tidepool program to patients who fit these criteria. The outgoing call/email will consist of questions to find out why the event happened and then suggestions on how to trouble shoot to avoid issues in the future. If needed the patient will be seen in person for an education/training session. If the patient cannot be reached within 6 hours, the patient's emergency contact will be notified if the PI feels that such out reach is warranted.

Visit 2 - will occur at 14 weeks. Questionnaires will be administered, A1C measured and CGM data and compare to baseline.

DATA COLLECTION AND TESTING PROCEDURES (Baseline, and 14 weeks) HbA1c - HbA1c will be obtained using the point of care Siemens DCA Vantage Analyzer.

Continuous Glucose Monitoring (CGM)- A commercially available DexCom G5 or G6 CGM device will be provided and a sensor will be inserted. The participant will receive instructions on calibration, insertions, maintenance, use, and removal of the sensor.

T1D REDEEM Diabetes Distress Questionnaire- The T1D REDEEM Diabetes Distress Questionnaire measures several dimensions of stress related to having type 1 diabetes. It consists of the following 7 subscales: Subscale 1 - Powerlessness (5 items); Subscale 2 - Management Distress (4 items); Subscale 3 - Hypoglycemia Distress (4 items); Subscale 4 - Negative Social Perceptions (4 items); Subscale 5 - Eating Distress (3 items); Subscale 6 - Physician Distress (4 items); Subscale 7 - Friend/Family Distress (4 items). Each question has a 6-choice Likert response format. Administration time is approximately 10 minutes.

Hypoglycemia Fear Survey - The Hypoglycemia Fear Survey measures several dimensions of fear of hypoglycemia among adults with type 1 diabetes. It consists of a 10-item Behavior subscale that measured behaviors involved in avoidance and over-treatment of hypoglycemia and a 13-item Worry subscale that measures anxiety and fear surrounding hypoglycemia, each with a 5-choice Likert response format. Administration time is approximately 10 minutes.

Simplified Diabetes Knowledge Test -The Simplified Diabetes Knowledge Test consists of 23 knowledge test items developed by the Michigan Diabetes Research Training Center (MDRTC). These items represent a test of general knowledge of diabetes and are answered in a true/false/don't know format. The psychometric properties provide information regarding the reliability of the various groups of items, as well as a difficulty index (percent of patients who scored this item correctly), and an item to group total correlation for each item. These data can be reported when describing the use of the test. Administration time is approximately 15 minutes.

Assessment of Sever Hypoglycemia and Diabetic Ketoacidosis -The Assessment of Severe Hypoglycemia and Diabetic Ketoacidosis is an interviewer administered survey assessing if the subject had any episodes of severe hypoglycemia and/or diabetic ketoacidosis since their last study visit. Events are recorded to assess frequency, as is type of assistance required to treat the event. Administration time is approximately 5 minutes.

TIDEPOOL. https://tidepool.org/ Tidepool is an open source, not-for-profit company focused on "liberating data from diabetes devices, supporting researchers, and providing free software to people with diabetes and their care teams." Tidepool is the program that is used routinely in our clinic to assess data from diabetes devices. As part of clinical care all patients are encouraged to upload their data to Tidepool for analysis. Currently we have over 250 patients streaming data into Tidepool. However, data is not analyzed on a daily basis, but rather on as "as needed" basis if a patient contacts the clinic with a problem.

Tidepool is an FDA registered entity. The software is listed with the FDA under regulations 880.6310 and 862.2120 as Class I/Exempt medical devices and Medical Data Display Systems. Tidepool complies with all applicable FDA regulations including 21 code of federal regulations (CFR) 820 Quality System Regulations. Class I/Exempt and medical device data system (MDDS) software are exempt from FDA part 510(k) filing and approval requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 diabetes
2. Age >65 years old
3. Insulin regimen involves either use of an insulin pump or multiple daily injections of insulin.
4. Understand the study requirements and agree to comply with all study visits and procedures, including the use of the study CGM.
5. Fluent in English or Spanish
6. Must have a smart phone

Exclusion Criteria:

1) No serious illnesses where life expectancy is <1 year

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
CGM-Tele-monitoring effects on hypoglycemia | 14 weeks
  Number of patients with lower incidents of hypoglycemia as assessed by CGM data and self report from baseline to 14 weeks.

SECONDARY OUTCOMES:
CGM-Tele-monitoring effects on CGM adherence | 14 weeks
  Number of patients with increased CGM use as assessed by number of days CGM data is available for download from baseline to 14 weeks.
CGM-Tele-monitoring effects on hypoglycemic fear | 14 weeks
  Number of patients with decreased hypoglycemic fear as measured by reduction in the hypoglycemic fear scale from baseline data to 14 weeks
CGM-Tele-monitoring effects on diabetes distress | 14 weeks
  Number of patients with decreased diabetes distress as measured by reduction in the diabetes distress scale from baseline data to 14 weeks.
CGM - Tele-monitoring effects on diabetes knowledge | 14 weeks
  Number of patients with increased diabetes knowledge as measured by an increase on the simplified diabetes knowledge test from baseline to 14 weeks.
CGM - Tele-monitoring effects on diabetic ketoacidosis | 14 weeks
  Number of patients with decreased incidents of diabetic ketoacidosis as measured by self-report from baseline to 14 weeks.
CGM - Tele-monitoring effects on HbA1c | 14 weeks
  Number of patients with decreased HbA1c as measured by point of care HbA1c level from baseline to 14 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Peters, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Westside Center for Diabetes, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/96/NCT04328896/Prot_000.pdf